CLINICAL TRIAL: NCT04332263
Title: Development and Application of a Portable Electrical Stimulator With Biofeedback to Increase Mobility and Improve the Neuromuscular Function of Critical Adult Patients in Intensive Care Units
Brief Title: Neuromuscular Electrical Stimulation in ICU Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the pandemic we were unable to recruit patients from the hospital
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, Full Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36588914.4.1001.5347
Record Dates: First submitted 2019-06-07; First posted 2020-04-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Intensive Care Unit Acquired Weakness

STUDY DESIGN:
Intervention Model Description: The present study is a randomized controlled trial, which followed the recommendations proposed by the CONSORT Statement
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized through data generated by a computer program containing the coded distribution (Randomizer, USA). The software takes into account one of the main objectives of randomization, which is to prevent the researcher from identifying which intervention will be performed on each patient. A researcher blinded to the study will do the generation of the sequence of numbers, after the patients' selection by the inclusion and exclusion criteria. The numbers sequence used for randomization will be kept confidential until the exact moment of the beginning of the intervention. In addition, a second blinded researcher, who will not be aware of the subjects' names in the three experimental groups, will perform the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Electrical Stimulation - NMES (Experimental): NMES will be applied bilaterally on the quadriceps femoris muscle of ICU patients. An electrical stimulation system and an ICU-designed dynamometer will be used with the patients lying in bed, with the hips and the knees flexed at 60 and 90 degrees, respectively. Supramaximal single-pulse's peak force will be used to determine the NMES intervention level. NMES (alternating biphasic current, stimulation frequency = 80 Hz, 1 ms pulse duration) will be used to evoke tetanic forces (EF) at 50% of the supra-maximal single-pulse EF (i.e., 10-12% of a maximal voluntary isometric contraction). NMES protocol will be performed five times a week, lasting 20 min. Muscle fatigue will be evaluated every 5 min of the intervention, and will be determined as a 10 % decrease in the single-pulse evoked torque between the evoked force produced pre- and during the NMES protocol. If and when a 10% reduction of the single-pulse EF is achieved, the intervention protocol will be terminated before the 20 min.
  Interventions: Other: Neuromuscular Electrical Stimulation - NMES
- Control Group - CG (No Intervention): The control group (CG) will only perform conventional physiotherapy and will not receive any NMES training, but will be evaluated through the same evaluations and in the same moments of the two above mentioned intervention groups. Conventional physiotherapy will be given to all three groups.

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation - NMES — NMES will be applied through an alternating biphasic current, with a stimulation frequency of 80 Hz and 1 ms pulse duration. Tetanic evoke forces (EF) at a 50% level of a supra-maximal single-pulse peak EF (i.e., 10-12% of a maximal voluntary isometric contraction) will be used. NMES protocol will be performed five times a week, lasting 20 minutes. Muscle fatigue will be evaluated every 5 min of the intervention, and will be used to determine the NMES protocol termination. A 10 % decrease in the single-pulse evoked torque between the evoked force produced pre- and during the NMES protocol will be used to terminate the fatigue protocol.
  Other Names: Artificial electrical stimulation
  Arms: Neuromuscular Electrical Stimulation - NMES

SUMMARY:
The aim of the present study is to evaluate the effects of neuromuscular electrical stimulation (NMES) combined with conventional physiotherapy (Experimental Group), compared to conventional physiotherapy only (Control Group) in critically ill Intensive Care Unit (ICU) patients, by means of a randomized controlled clinical trial. The investigators expect that the NMES program will be able to reduce muscle structure and function losses compared to control group, and will improve muscle quality faster, will reduce the ventilation time and the total time spent at the ICU, as well as improve functionality of these patients. In addition, the researchers expect to understand which mechanisms determine such adaptations in the musculoskeletal system of these patients.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the effects of neuromuscular electrical stimulation (NMES) combined with conventional physiotherapy (Experimental Group), compared to conventional physiotherapy only (Control Group) in critically ill ICU patients, by means of a randomized controlled clinical trial. Primary outcomes evaluated during ICU patient's hospitalization are (1) the time spent in the ICU; (2) time of mechanical ventilation; (3) time and success of weaning (up to 48 hours), (4) the isometric torque from contractions artificially generated by NMES and evaluated by dynamometry; (5) muscle morphology and quality by means of ultrasonography. Secondary outcomes include (6) the sit and stand test; (7) gait speed test; (8) autonomic control (heart rate variability); (9) peripheral polyneuropathy by means of MRC scale; (10) Inflammatory profile - inflammatory (IL-6 and TNF-α) and anti-inflammatory (IL-10) cytokines; (11) blood muscular biochemical markers (IGF1, LDH, CK); (12) predictive mortality index for patients admitted to the ICU (SAPS 3); (13) survival rate; and (14) mobility (PERME). After discharge from the ICU or as soon as the patients are able to perform force voluntarily, the maximum voluntary torque will also be evaluated by means of dynamometry. Also, clinical data, hemodynamic variables, dosage of neuromuscular blockers and corticosteroids, blood glucose levels in the morning, daily water balance, oxygenation index, arterial blood gases, mechanical ventilator parameters, Glasgow scale, sedation scale (RASS), will be recorded daily. The investigators expect that the NMES program will be able to reduce muscle structure and function losses compared to control group, and will improve muscle quality, will reduce the ventilation time and the total time spent at the ICU, as well as improve functionality of these patients. In addition, the researchers expect to understand which mechanisms determine such adaptations in the musculoskeletal system of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any clinical condition hospitalized in the ICU, which are monitored by the Physiotherapy Service:
* Cerebrovascular diseases
* Other bacterial diseases
* Circulatory and respiratory diseases
* Digestive and abdominal diseases
* Liver diseases
* Time between the patient's ICU entry and the onset of the NMES intervention less than one week.

Patients may be in mechanical ventilation, non-invasive ventilation, oxygen therapy or oxygen ambient ventilation (no ventilatory add). Patients re-admitted to the ICU within the same hospitalization period (i.e., did not leave the hospital) may also be included, as well as patients with previous tracheostomy.

Exclusion Criteria:

* Previously diagnosed neuromuscular diseases:
* ALS
* Guillain Barre
* Chronic stroke
* TRM
* End-stage malignant disease
* Lower limbs' amputation
* Body mass index above 40 kg/m2
* Cachexia (defined as the presence of chronic disease and weight loss ≥ 5% in a period shorter than 12 months or BMI < 20 kg/m2, associated with at least three of the following criteria: (1) decreased muscle strength; (2) fatigue; (3) anorexia; (4) reduction of fat free mass index; and (5) biochemical abnormalities such as inflammation, anemia or reduction of serum albumin concentration).
* Lesions on the skin at the electrode placement and/or dynamometer support points
* Post-operative transplantation
* Patients using a neuromuscular blocker
* Hemodynamic instability (nora > 10; ABCDE criteria)
* Height < 1.50m
* Rhabdomyolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Total ICU time | Immediately after each patient discharge from the ICU (7 to 15 days after entry at the ICU, on average).
  Total time of stay at the ICU, from admission to discharge (an average of 7 up to 15 days). Total ICU time will be collected from the patient's medical record.
Mechanical ventilation time | Immediately after each patient mechanical ventilation release (2 to 5 days from intubation start, on average).
  Total time of mechanical ventilation, from patient intubation to weaning, will be collected from the patient's medical record.
Weaning time | Immediately after each patient discharge from the ICU (7 to 15 days after entry at the ICU, on average).
  Time and success of weaning post-mechanical ventilation, from weaning to ICU discharge, will be collected from the medical record of the patient. The maintenance of spontaneous ventilation for at least 48 hours after discontinuation of artificial ventilation will be considered a successful weaning.
Change in knee extensor evoked force | Change from the patient ICU admission to immediately before ICU discharge (e.g., from day 1 to day 7-15, on average).
  Knee extensor evoked force (EF) will be evaluated by means of isometric tests using a stainless steel dynamometry system instrumented with a load cell. EF will be evaluated through evoked contractions of the knee extensor muscles generated by supramaximal electrical stimuli with symmetrical rectangular biphasic current, applied in the form of single pulses (phase duration=1 ms, pulse duration=2 ms). At the beginning of the tests, the singular pulses will be applied with a manual trigger, and current intensity will be gradually increased (maximum 180 mA, inter-pulse interval = 3-5 second), until no further EF increase is observed. The current intensity required to reach the peak EF will then be increased by 10% to ensure supra-maximal stimulus during the tests. Three singular pulses will be applied and EF will be obtained by the mean value from the three evoked contractions. The change in knee extensor EF will be calculated as the difference in EF from ICU admission to ICU discharge.
Knee extensor maximal voluntary isometric contraction | Immediately before each patient ICU discharge (7 to 15 days after admission, on average).
  Maximal knee extensor strength capacity during voluntary effort will be assessed only when the patient is discharged (POST) from ICU, by performing maximum voluntary isometric contractions (MVICs). To do so, once properly positioned on the dynamometer, subjects will perform three knee extensor MVICs, maintaining each contraction for a 5 sec period each. Subjects will be instructed to perform the contractions without any visual feedback, rapidly increasing the effort until they reach the maximum torque production, which should be maintained until the verbal command to cease contraction. Two-minute intervals will be given between contractions. The highest torque value recorded during the three MVICs will be adopted as the maximum voluntary effort (maximal torque). Mean and standard deviation values from the MVICs will be calculated for the experimental groups.
Knee extensor muscle quality: Real-time ultrasound 9 MHz frequency | Immediately after each patient ICU admission and immediately before ICU discharge (7 to 15 days on average).
  Real-time ultrasound (Vivid-I, General Electric, USA) obtained with a linear array probe (4 cm wide) and a 9 MHz sampling frequency will be used for the evaluation of muscle quality. Images from the rectus femoris (RF) muscle will be obtained with the participants at rest. Ultrasound images will be captured in the muscle's transverse plane, at 50% of the muscle's belly. To ensure the ultrasound images comparison at different times, the brightness and contrast settings will be maintained at 50% during all evaluations. Muscle quality will be determined using a standard function of the Image-J (National Institute of Health, USA) software. A region of interest that includes as much muscle area as possible, avoiding the fascia, will be selected from the RF muscle images. Muscle quality will be determined by analysing the image's average gray scale, which ranges from total black (0) to total white (255), and mean values from three ultrasound images will be determined.
Rectus femoris cross-sectional area | Immediately after each patient ICU admission and immediately before ICU discharge (7 to 15 days on average).
  RF cross-sectional area (CSA) will be captured at rest in the muscle's transverse plane, at 70% of the muscle belly. The probe will be positioned transversely to the muscle belly, with the image depth adjusted so that both the RF superficial and deep aponeuroses can be visualized. RF CSA will be obtained through the analysis of these transverse images. A standard function of the Image-J (National Institute of Health, USA) software will be used, which allows the demarcation of the muscular perimeter (excluding the aponeuroses), and calculates the internal selected area (cm2). The mean CSA value from three images will be calculated for each group at each time-point of the study.
Knee extensors muscle thickness | Immediately after each patient ICU admission and immediately before ICU discharge (7 to 15 days on average).
  Muscle thickness (MT) will be obtained at rest from ultrasound images of the RF, vastus intermedius (VI), vastus lateralis (VL) and vastus medialis (VM) muscles. Ultrasound images will be captured at 50% of the RF, VI and VL muscle bellies, and at 70% of the VM length. MT will be obtained by image analysis in the Image-J software (National Institute of Health, USA). Five equidistant measurements will be taken from the superficial to deep aponeurosis of the VI, VL and VM muscles. RF diameter will be obtained from the transverse image obtained for muscle quality evaluation and will represent its MT. The mean value of the five measures of the VI, VL and VM muscles will be calculated for each image. The mean MT value from three ultrasound images will be calculated and will be used as the MT from each evaluated muscle (in cm).

SECONDARY OUTCOMES:
Sit to stand test | Immediately after each patient ICU discharge (7 to 15 days after admission, on average).
  The sit to stand test measures the total time required to perform 5 repetitions of the sit to stand movement on a chair. The test begins with the participant sitting on a chair with trunk support, feet at a shoulder-width apart, and fully resting on the ground. The upper limbs will be crossed at chest height. At the "start signal", the participant moves to the standing position, rising to the upright position (vertical position), and next returning to the initial sitting position. The test results will consist of assessing the total time taken by the patient to perform five repetitions of the movement of getting up and sitting down on the chair as quickly as possible.
Waking Speed Test | Immediately after each patient ICU discharge, until study completion (about 30 months).
  The Walking Speed Test will be performed in a flat corridor, in which the patient is asked to walk as fast as possible a 10-meter distance previously marked on the ground. The travel time in the central 6 meters of the 10-meter distance will be measured. Running speed ≤ 0.8 m/s will be considered as low physical performance. Patients will be familiarized with the test by the evaluator simulating the test performance prior to the test.
Heart rate variability | Immediately before and during NMES intervention protocols (daily, from 7 to 15 days on average).
  Heart rate variability (HRV) will be evaluated by recording the heart rate at the beginning of the tests, at the second half of a 10-min rest for HRV baseline values assessment. After that, HRV will be obtained during the NMES protocols. HRV records will be obtained with a Polar heart rate monitor (POLAR RS800CX, USA) that will be placed on the subjects' precordium region. Data analysis will be performed by studying the heartbeats RR intervals imported into Kubios software (version 3.0.2, Finland). Analyzes will be performed in the domains of (1) time, by means of both the mean heart rate (beats/min) and the mean values of the intervals between the R-waves (ms); and (2) frequency, by calculating both the spectral power values of the low frequency (LF) and high frequency (HF) components (normalized unit; n.u.). Five-minute windows will be analyzed, obtained from the second half of the REST period just before the tests, and 5 min within the second half of the NMES protocol.
Peripheral polyneuropathy | Immediately before ICU discharge (7 to 15 days after admission, on average).
  Peripheral polyneuropathy will be assessed through the MRC (Medical Research Council) scale. Three muscle groups in all four limbs will be evaluated through this scale, with values ranging from 0 (quadriplegia) to 60 points (normal muscle strength). The following functions will be evaluated: wrist flexion, forearm flexion, abduction of the shoulder, ankle dorsiflexion, knee extension and hip flexion. Patients with a score lower than 48 out of 60 points will be diagnosed with peripheral polyneuropathy.
Inflammatory profile | Immediately after each patient ICU admission and immediately before ICU discharge (7 to 15 days on average).
  Immunological reagents will be used to detect anti and pro-inflammatory cytokines. The serum production of IL-6, IL-10 and TNF-α will be determined by ELISA.
Muscular biochemical markers | Immediately after each patient ICU admission and immediately before ICU discharge (7 to 15 days on average).
  The IGF1, creatine kinase and phosphocreatine markers will be analyzed from blood collection in a serum tube with EDTA. The blood will be centrifuged in refrigerated medium for 15 minutes at 3000g and the plasma will be stored separately in a freezer at -80°C for analysis of these markers.
Mobility (PERME) | Immediately before each patient ICU discharge (7 to 15 days after admission, on average).
  This instrument comprises 15 items grouped into 7 categories (scored from 0 to 32 points in total): (1) mental state, which evaluates the ability of patients to obey commands; (2) potential barriers to mobility, which verifies the presence of devices that can impede mobility; (3) strength, which evaluates the ability to perform both hip flexion above 20º with extended knee, as well as shoulder flexion above 45º with elbows extended; (4) in bed mobility, which refers to the ability to transfer from dorsal decubitus to the seated position, and maintenance of the seated position at the bedside; (5) transfers, which refers to the ability to transfer from sitting to standing, orthostatism and transfer from the bed to the armchair are evaluated; (6) gait, which is assessed as the ability to walk (or not) with severe, moderate or little assistance; (7) endurance, which is the ability to walk a certain amount of steps in 2 minutes. In this instrument, a high score indicates high mobility.
Arterial pressure | Daily from ICU admission to discharge day (7 to 15 days on average).
  Systemic arterial pressure (mmHg) and mean arterial pressure (mmHg), collected from medical records.
Heart rate | Daily from ICU admission to discharge day (7 to 15 days on average).
  Mean heart rate (bpm), collected from medical records.
Ventilatory mode | Daily from ICU admission to discharge day (7 to 15 days on average).
  Ventilatory mode (PCV, VCV, PSV), collected from medical records.
Tidal volume | Daily from ICU admission to discharge day (7 to 15 days on average).
  Tidal volume (ml), collected from medical records.
Ventilator frequency | Daily from ICU admission to discharge day (7 to 15 days on average).
  Ventilator frequency (rpm), collected from medical records.
Sensitivity | Daily from ICU admission to discharge day (7 to 15 days on average).
  Sensitivity (cmH2O or L/min), collected from medical records.
FiO2 | Daily from ICU admission to discharge day (7 to 15 days on average).
  FiO2 (%), collected from medical records.
PEEP | Daily from ICU admission to discharge day (7 to 15 days on average).
  PEEP (cmH2O), collected from medical records.
Water balance | Daily from ICU admission to discharge day (7 to 15 days on average).
  Water balance (mL), collected from medical records.
Oxygenation rate | Daily from ICU admission to discharge day (7 to 15 days on average).
  Oxygenation rate (PaO2 / FiO2 ratio), collected from medical records.
Arterial blood gas analysis | Daily from ICU admission to discharge day (7 to 15 days on average).
  PaCO2 (mmHg), PaO2 (mmHg) and HCO3- (mEq/L), collected from medical records.
Glasgow scale | Daily from ICU admission to discharge day (7 to 15 days on average).
  Glasgow scale (range 3-15), collected from medical records.
RAMSAY scale | Daily from ICU admission to discharge day (7 to 15 days on average).
  RAMSAY scale (range -5 to +4), collected from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil